CLINICAL TRIAL: NCT04801667
Title: Prospective Study in a Single Center to Evaluate the Impact, Safety, Tolerability and Immunogenicity of the Coronavac Vaccine in Kidney Transplant Recipients
Brief Title: Evaluate the Impact, Safety, Tolerability and Immunogenicity of the Coronavac Vaccine in Kidney Transplant Recipients
Acronym: TXCoronavac
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital do Rim e Hipertensão (Other)
Responsible Party: Principal Investigator, Helio Tedesco Silva Junior, Affiliate teacher, Hospital do Rim e Hipertensão
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TxR Coronavac - Hrim
Record Dates: First submitted 2021-03-10; First posted 2021-03-17 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: SARS-CoV Infection; Coronavirus Infection; Vaccine Adverse Reaction
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Coronavirus Infections | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronavac vaccine (Experimental): Kidney transplant recipients receiving the coronavac vaccine
  Interventions: Biological: Coronavac

INTERVENTIONS:
Biological: Coronavac — The CoronaVac is manufactured by Sinovac Life Sciences Co., Ltd. This vaccine contains the inactivated SARS-CoV-2 virus antigen and is administered intramuscularly.

SUMMARY:
Since the beginning of the SARS-CoV-2 pandemic, 1031 (8.7%) of the 11875 kidney transplant recipients being followed up at Hospital do Rim have been infected. The overall lethality rate was 24%, reaching 53% among those over 70 years old. Among the survivors, there is also a high incidence of renal dysfunction with loss of the renal graft and definitive return to dialysis. Patients receiving pharmacological immunosuppression, including transplant recipients, have not been included in the studies carried out to date. In addition, kidney transplant recipients may have reduced vaccine responses compared to the general population. The severity, the high incidence of renal dysfunction and loss of renal graft, and the high lethality associated with COVD-19 justify the investigation of the epidemiological impact and immunogenicity of the vaccine against SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 18 years old;
2. Time after transplantation greater than 3 months;
3. Time after treatment with anti-thymocyte globulin longer than 4 weeks;
4. Able and willing (in the investigator's opinion) to comply with all study requirements;
5. Provide written informed consent

Exclusion Criteria:

1. Planned receipt of any vaccine (authorized or experimental), within 30 days before and after vaccination;
2. Prior receipt of an experimental or authorized vaccine with the possibility of impacting the interpretation of the study data (for example, vectorized vaccines by Adenovirus, any vaccines against coronavirus);
3. Administration of immunoglobulins and / or any blood products in the three months prior to the planned administration of the candidate vaccine;
4. Any history of angioedema or anaphylaxis;
5. Pregnancy, lactation or willingness / intention to become pregnant during the study;
6. Diagnosis or current treatment for cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ);
7. History of severe psychiatric illness that possibly affects your participation in the study;
8. Hemorrhagic disorder (eg, factor deficiency, coagulopathy or platelet disorder) or a previous history of significant bleeding or hematoma after IM injections or venipuncture;
9. Continued use of anticoagulants, such as coumarins and related anticoagulants (for example, warfarin) or new oral anticoagulants (for example, apixaban, rivaroxaban, dabigatran and edoxaban);
10. Current suspected or known addiction to alcohol or drugs.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3371 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence of hospitalization or death in 28 days associated with COVID-19 (symptomatic cases confirmed virologically by COVID -19 with positive CRP) 14 ± 2 days after the second dose of the vaccine. | 45 days

SECONDARY OUTCOMES:
Evaluate the impact of the vaccine on the incidence of COVID-19 according to the severity criterion of the World Health Organization. | 6 months
Evaluate the impact of the vaccine on the incidence of COVID-19 and hospitalization for COVID-19 disease, confirmed by PCR, for a period of 6 months after the final vaccination. | 6 months
Evaluate the vaccine's safety, tolerability, and reactogenicity profile: occurrence of signs and symptoms of local and systemic reactogenicity requested seven days after vaccination. | 7 days
Evaluate the incidence of serious adverse events for a period of 6 months after the final vaccination. | 6 months
Evaluate immunogenicity by detecting antibodies against SARS-CoV-2 for a period of 6 months after the final vaccination. | 6 months
  IgG antibody levels will be used to assess immunogenicity.
Analysis of the genetic sequencing of SARS-CoV-2 in patients who test positive for SARS-CoV-2 PCR. | 6 months
  Genetic sequencing of the virus will be carried out, that is, reading the genome of Sars-Cov-2, to evaluate possible new variants.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital do Rim - Fundação Oswaldo Ramos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Medina-Pestana J, Covas DT, Viana LA, Dreige YC, Requiao-Moura LR, Nakamura MR, Lucena EF, Foresto RD, Tedesco-Silva H, Cristelli MP. Homologous Third Dose of Inactivated Whole-virion Vaccine Fails to Elicit a Robust Immune Response Among Kidney Seronegative Transplant Recipients. Transplantation. 2022 May 1;106(5):e284-e285. doi: 10.1097/TP.0000000000004029. Epub 2021 Dec 28. No abstract available. PMID 34974453
- [Derived] Medina-Pestana J, Covas DT, Viana LA, Dreige YC, Nakamura MR, Lucena EF, Requiao-Moura LR, Fortaleza CMCB, Foresto RD, Tedesco-Silva H, Cristelli MP. Inactivated Whole-virus Vaccine Triggers Low Response Against SARS-CoV-2 Infection Among Renal Transplant Patients: Prospective Phase 4 Study Results. Transplantation. 2022 Apr 1;106(4):853-861. doi: 10.1097/TP.0000000000004036. PMID 34882589
- [Derived] Medina-Pestana J, Cristelli MP, Viana LA, Foresto RD, Requiao-Moura LR, Tedesco-Silva H, Covas DT. Clinical Impact, Reactogenicity, and Immunogenicity After the First CoronaVac Dose in Kidney Transplant Recipients. Transplantation. 2022 Jan 1;106(1):e95-e97. doi: 10.1097/TP.0000000000003901. No abstract available. PMID 34292214